CLINICAL TRIAL: NCT05237466
Title: Motivational Interviewing to Enhance Behavioral Change in Older Adults with Hoarding Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mississippi State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mary Dozier, Assistant Professor, Mississippi State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-561; 1R15MH127565-01A1 (NIH)
Record Dates: First submitted 2022-01-14; First posted 2022-02-14 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Hoarding Disorder
MeSH Terms: conditions — Hoarding Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RECLAIM: Reducing Clutter and Increasing Meaning (Experimental): Participants will receive a combination of motivational interviewing and sorting practice to reduce hoarding symptoms.
  Interventions: Behavioral: RECLAIM: Reducing Clutter and Increasing Meaning
- Sorting Practice (Active Comparator): Participants will receive sorting practice only to reduce hoarding symptoms.
  Interventions: Behavioral: Sorting Practice

INTERVENTIONS:
Behavioral: RECLAIM: Reducing Clutter and Increasing Meaning — Participants will receive 16 weekly 1-hour treatment sessions in their home delivered by Masters-level clinicians with the assistance of undergraduate researchers. Each treatment session will involve a combination of motivational interviewing (MI) and sorting practice. The rationale behind the sorting practice is to develop the skill of sorting and the formation of a daily sorting routine. The MI portion of the initial session will involve an evaluation of client strengths and individual biopsychosocial goals. The initial and subsequent sessions will include a variety of MI techniques, including decisional balancing, developing discrepancy, personalized feedback, and reinforcement of responsibility of sense of self-efficacy.
  Arms: RECLAIM: Reducing Clutter and Increasing Meaning
Behavioral: Sorting Practice — Participants will receive 16 weekly 1-hour treatment sessions in their home delivered by Masters-level clinicians with the assistance of undergraduate researchers. Clinicians will encourage participants to sort objects during each session while refraining from use of any specific cognitive or motivational therapeutic techniques. Participants will be asked to record the frequency and duration of any sorting/ discarding they did during the previous week.
  Arms: Sorting Practice

SUMMARY:
This study will compare two behavioral interventions for hoarding disorder in older adults.

DETAILED DESCRIPTION:
Hoarding disorder is a psychological condition with a unique constellation of consequences for older adults, including increased risk of fire and dying in a fire, insect infestation, and medical problems. Dangers related to cluttered living spaces are exacerbated by reduced executive functioning, attention, and concentration. Hoarding psychopathology results from maladaptive cognitions (e.g., desire to keep items others would discard) and maladaptive behavioral patterns (e.g., avoidance of sorting/discarding items).

Extant treatments for hoarding have targeted fear reduction as the mechanism of change, either through cognitive-behavioral therapy focusing on cognitive restructuring or behavior therapy focusing on exposure therapy. Older adults have a lackluster response to cognitive restructuring for hoarding, and, although exposure therapy increases treatment response, both approaches require a lengthy six-month dose. Our preliminary work suggests that fear reduction may not be a universally relevant target mechanism for older adults, and that to be responsive to the specific needs of older adults, other mechanisms need to be identified.

Motivational interviewing is a technique that is already typically incorporated into hoarding treatment and has been demonstrated to increase motivation for behavioral change across a range of health conditions for older adults, including physical activity, diet, and disease management. Because sorting/discarding is at its core a health behavior that hoarding patients lack the motivation to engage in, motivational interviewing is likely to decrease hoarding severity by eliciting increased levels of sorting/discarding.

The proposed project will use a mechanistic clinical trials approach to determine if a four-month intervention combining motivational interviewing with sorting practice can engage the proposed target, motivation for behavioral change, when compared to a four-month dose of sorting practice alone in a sample of rural-dwelling older adults with hoarding disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60+
* Live within a 60-minute driving radius of Starkville, MS
* Have a primary psychiatric diagnosis of hoarding disorder

Exclusion Criteria:

* Major cognitive impairment
* Active psychosis, drug use, or acute suicidal ideation
* Concurrent psychotherapy focused on hoarding
* Changed psychotropic medications within the past three months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of sorting/discarding behavior | Four months
  As a behavioral indicator of motivation to engage in sorting/discarding behavior, participants will be asked to report at baseline and at their weekly treatment sessions the frequency of sorting/discarding items in the previous week.
Change in duration of sorting/discarding behavior | Four months
  As a behavioral indicator of motivation to engage in sorting/discarding behavior, participants will be asked to report at baseline and at their weekly treatment sessions the duration of sorting/discarding items in the previous week.
Change in score on the University of Rhode Island Change Assessment Questionnaire McConnaughy et al., 1983) | Four months
  The URICA is a 32-item Likert scale that assesses readiness for change and includes four subscales that individually assess stage of change (Precontemplation, Contemplation, Action, and Maintenance). Previous investigations have found adequate internal reliability for the URICA in treatment-seeking samples (Dozois et al., 2004), including in older hoarding samples specifically (Ayers et al., 2019).
Change in score on the Apathy Evaluation Scale (AES-S; Marin, 1991) | Four months
  The AES is an 18-item measure of an individual's deficits in goal-directed thoughts and behavior. The AES was developed specifically to assess apathy in adults aged 55+ and is predictive of motivation for behavioral change (Resnick et al., 2012).

SECONDARY OUTCOMES:
Rating on the Treatment Acceptability/ Adherence Scale (TAAS; Milsevic et al., 2015) | Immediately after session one
  The TAAS is a 10-item self-report measure of a patient's perception of the acceptability of a treatment as well as their anticipated adherence to the protocol.

OTHER OUTCOMES:
Change in score on the Saving Inventory-Revised (SI-R; Frost et al., 2004) | Four months
  The SI-R is a 23-item measure of the three core hoarding symptoms (urges to save, difficulty discarding, and excessive clutter).
Change in score on the Clutter Image Rating (CIR; Frost et al., 2008) | Four months
  The CIR is a three-item pictorial rating scale of clutter level in the bedroom, kitchen, and living room. Assessor ratings of the CIR will be used for the proposed project.
Change in scores on the Behavioral Approach Task for sorting/discarding(BAT; Dozier & Ayers, 2017; Dozier et al., 2020) | Four months
  The BAT involves the participant sorting items in a cluttered part of their home for 15 minutes. The speed of sorting and percentage of items discarded will be used as behavioral indicators of hoarding severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Mississippi State University, Starkville, Mississippi, United States

IPD SHARING:
Plan to Share IPD: Yes
All data collected will be shared using the NIMH Data Archive (NDA) following safe harbor requirements for de-identification. Data dictionaries currently available in NDA will be used for most measures assessed (e.g., PROMIS measures), but new data dictionaries will be created for unique data elements (e.g., reported frequency of sorting behavior) and standardized measures not currently entered in the NDA (e.g., Clutter Image Rating). Data will be deposited in the NDA twice per year over the course of the study and once the study is complete. Each manuscript based off the study will have specific analytic files deposited to the NDA once the manuscript is accepted for publication.